CLINICAL TRIAL: NCT02297503
Title: An Evaluator-blinded Multi-center Study of Combined Treatment With Azzalure, Restylane/Emervel Filler and Restylane Skinbooster as Compared to Single Treatment With Either Azzalure Alone or Restylane/Emervel Filler Alone
Brief Title: Safety and Efficacy of Treatment With Azzalure, Restylane/Emervel Filler and Restylane Skinbooster
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1211
Record Dates: First submitted 2014-10-31; First posted 2014-11-21 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-08

CONDITIONS: Facial Aesthetic Treatment
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azzalure alone as single treatment (Experimental): Azzalure alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
  Interventions: Drug: Azzalure; Device: Restylane/Emervel filler; Device: Restylane Skinbooster
- Filler alone as single treatment (Experimental): HA filler alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
  Interventions: Drug: Azzalure; Device: Restylane/Emervel filler; Device: Restylane Skinbooster

INTERVENTIONS:
Drug: Azzalure — Glabellar lines
  Other Names: Botulinum toxin
Device: Restylane/Emervel filler — Facial tissue augmentation
  Other Names: Hyaluronic acid
Device: Restylane Skinbooster — Facial skin rejuvenation
  Other Names: Hyaluronic acid

SUMMARY:
The efficacy and safety, as well as subject satisfaction will be evaluated after single treatment with Azzalure alone or Restylane/Emervel filler alone followed by repeated combined treatment with Azzalure, Restylane/Emervel filler and Restylane Skinbooster. Subjects will be followed for up to 18 months after initial treatment.

ELIGIBILITY:
Inclusion Criteria

* Subjects aged 35 to 50 years old
* Subjects with the intention to undergo facial aesthetic treatment and who are likely to benefit from a combination of injection treatments and the benefit can be shown by improvements in their global facial aesthetic appearance and satisfaction.
* Subjects with nasolabial folds assessed as mild or moderate.
* Subjects with glabellar lines assessed as moderate or severe, when the severity of the lines has an important psychological impact on the subject.
* Subjects with signed informed consent.

Exclusion Criteria:

* Subjects requiring treatment of forehead lines or crow´s feet.
* Obvious facial sagging (major loss of facial fat/volume).
* Signs or symptoms of eyelid ptosis or signs of compensatory frontalis muscle activity.
* Heavily scarred or sun-damaged facial skin.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster/herpes simplex near or on the areas to be treated.
* Cancerous or pre-cancerous lesions in the areas to be treated.
* Facial tissue augmenting therapy or revitalization treatment with hyaluronic acid (HA) or collagen, or botulinum toxin treatment during the last 12 months.
* Procedures or treatments inducing an active dermal response such as laser, Intense Pulsed Light, chemical peeling, microdermabrasion, retinoids within the last 6 months.
* Any aesthetic surgery of the face.
* Permanent implant or aesthetic treatment with non-HA or non-collagen products in the face.
* History of severe keloids and/or hypertrophic scars.
* Neuromuscular junctional disorders (e.g. myasthenia gravis, Eaton Lambert syndrome or amyotrophic lateral sclerosis) or history of dysphagia and aspiration.
* Known hypersensitivity to hyaluronic acid, botulinum toxin, lidocaine hydrochloride or other amide-type anesthetics.
* History of autoimmune diseases.
* Any medical condition that in the opinion of the investigator would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may affect the general condition or may require frequent medical treatment).
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation (e.g. aspirin or other nonsteroidal anti-inflammatory drugs [NSAIDs]), Omega-3 or vitamin E within 10 days before study treatment, or a history of bleeding disorders.
* Immunosuppressive therapy, chemotherapy, or systemic corticosteroids within the last 3 months prior to baseline visit.
* Female subjects who are pregnant or plan to become pregnant within the study timeframe, or who are nursing.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kestemont, MD, Principal Investigator — Clinique Science et Beauté, Antibes, France
Locations (3):
- France (2):
  - Mediti Center, Paris, Antibes
  - Centre Medical Saint-Jean, Arras
- Akademikliniken, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Azzalure Alone as Initial Treatment: Azzalure alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
- Filler Alone as Initial Treatment: HA filler alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
Period: Overall Study
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Started | 30 | 31
Initial Single Treatment | 29 | 31
First Combined Treatment | 28 | 28
Second Combined Treatment | 28 | 28
Completed | 28 | 27
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Medical reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant withdrew consent after randomization and prior to first treatment. That participant is not included in the analyses.
Groups:
- Azzalure Alone as Initial Treatment: Azzalulre alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
- Filler Alone as Initial Treatment: Filler alone as single treatment at initial treatment followed by two combined treatments with Azzalure, HA filler and Skinboosters at Month 6 and Month 12.
- Total: Total of all reporting groups
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Full Range); unit: years] | 45.9 [36 to 50] | 43.6 [36 to 49] | 44.7 [36 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data on ethnicity only collected for the Swedish site.
  Participants
    White: number analyzed (Participants) | 11 | 11 | 22
    White | 11 | 11 | 22
Smoking [Number; unit: participants]
  Smoker | 9 | 10 | 19
  Non smoker | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Improvement in Global Facial Aesthetic Appearance at 7 Months (Review of Photographs)
Description: To evaluate "Global facial aesthetic appearance" at 7 months compared to at 1 month, blinded evaluator review of photographs.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Groups:
- Azzalure Alone as Initial Treatment: Subjects receiving Azzalure as initial treatment
- Filler Alone as Initial Treatment: Subjects receiving HA filler as initial treatment.
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 27 | 27
Participants | 20 | 25

2. Secondary Outcome: Number of Subjects With Improvement in Global Facial Aesthetic Appearance at 1, 7 and 13 Months (Review of Photographs)
Description: To evaluate "Global facial aesthetic appearance" at 1, 7 and 13 months, blinded evaluator review of photographs from the respective visits.
Time Frame: 1, 7 and 13 months
Population: Incorrectly taken photographs for six participants were excluded from analysis. Additionally two participants excluded because they were assessed different by all three evaluators.
Measure: Count of Participants; unit: Participants
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 23 | 25
Participants
  Superior Month 1 | 5 | 0
  Superior Month 7 | 5 | 11
  Superior Month 13 | 13 | 14

3. Secondary Outcome: Number of Participants Improved on the Global Aesthetic Improvement Scale (GAIS) as Assessed by Blinded Evaluator
Description: The 5-graded GAIS is used to assess the facial aesthetic improvement from baseline by responding to the question: "How would you describe the subject's global facial aesthetic appearance, compared to the photographs taken before treatment at baseline?" The scale grades are Very much improved, Much improved, Somewhat improved, No change, Worse. Improved subjects are those graded as Very much improved, Much improved, and Somewhat improved.
Time Frame: Month 1, Month 7, and Month 13
Population: Number of analyzed subjects decreased over time due to drop-out of study subjects.
  Data not presented "Per Arm", since statistical analysis was only performed on both groups combined after the combination treatments (since the groups receive the exact same treatment during the combination treatment).
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 60
participants
  Improved Month 1 | 35
  Improved Month 7: number analyzed (Participants) | 55
  Improved Month 7 | 42
  Improved Month 13: number analyzed (Participants) | 52
  Improved Month 13 | 47

4. Secondary Outcome: Number of Subjects Satisfied With Overall Facial Appearance (Questionnaire)
Description: Subjects answered the question "How satisfied are you today with the appearance of your face?" with "Very/somewhat satisfied", "Neither/nor", or "Very/somewhat dissatisfied". Number of subjects satisfied are those that answered "Very/somewhat satisfied".
Time Frame: Month 7 and Month 13
Measure: Number; unit: participants
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 28 | 28
participants
  Satisfied Month 7 | 23 | 26
  Satisfied Month 13 | 24 | 27

5. Secondary Outcome: Number of Subjects for Which the Investigator is Satisfied With Overall Facial Aesthetic Outcome
Description: The Investigator answered the question "How satisfied are you with the overall facial aesthetic outcome for the subject?" with "Very/somewhat satisfied", "Neither/nor", or "Very/somewhat dissatisfied". Satisfied criteria is met for those subjects that the Investigator answered "Very/somewhat satisfied".
Time Frame: Month 7 and Month 13
Measure: Number; unit: participants
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 28 | 28
participants
  Satisfied Month 7 | 28 | 28
  Satisfied Month 13 | 28 | 28

6. Secondary Outcome: Number of Participants Who Had Improvement in Wrinkle Severity Score of Treated Glabellar Lines (Validated Photo Scales)
Description: The wrinkle severity of the glabellar lines at maximum frown was evaluated by the investigator at baseline before first treatment and at follow-up visits. Validated photonumeric grading scales were used where each severity grade is illustrated by a set of photographs. The investigator performed the assessment live or by using 2D photographs from the present visit, together with the respective photo guide: 0 No glabella lines, 1 Mild glabella lines, 2 Moderate glabella lines, 3 Severe glabella lines, 4 Very severe glabella lines. Improved criteria is thus fulfilled for subjects receiving a lower score compared to baseline.
Time Frame: Month 7 and Month 13
Measure: Number; unit: participants
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 28 | 28
participants
  Improved Month 7 | 27 | 28
  Improved Month 13 | 27 | 28

7. Secondary Outcome: Change in Perceived Age of Subjects
Description: To evaluate First impression and perceived age of subjects by evaluation of photos.
  Change between timepoints are reported. A negative value indicates that the participant is assessed to be younger at the specified visit compared to the assessment made at 1 month after single treatment.
Time Frame: 1 and 7 months, and 1 and 13 months
Population: Five participants excluded from analysis due to incorrectly taken photographs.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 27 | 28
years
  Difference Month 7/Month 1 | -1.7 (4.0) | -1.9 (2.9)
  Differerence Month 13/Month 1: number analyzed (Participants) | 26 | 26
  Differerence Month 13/Month 1 | -1.9 (4.7) | -2.4 (2.9)

8. Secondary Outcome: Injected Filler Volume
Description: To evaluate the filler volume injected at initial single treatment and at following repeated combined treatment
Time Frame: Initial single treatment (baseline), first combined treatment (Month 6), and second combined treatment (Month 12)
Population: For the initial single treatment, only the "Filler alone as initial treatment" participants received filler. At the two combination treatments, all subjects received filler. Data from the "Filler alone as initial treatment" participants are presented for the single treatment while data for all subjects are presented for the combination treatments.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Filler Alone as Initial Treatment: The participants randomized to receive filler alone as initial single treatment.
- All Subjects: All subjects received filler at the combined treatments.
Arm/Group | Filler Alone as Initial Treatment | All Subjects
Number analyzed (Participants) | 31 | 56
mL
  Single and first combined treatment | 0.98 (0.06) | 1.92 (0.23)
  Second combined treatment: number analyzed (Participants) | 0 | 55
  Second combined treatment |  | 1.72 (0.50)

9. Secondary Outcome: Adverse Event Reporting
Description: To evaluate safety throughout the study period
Time Frame: 0-18 months
Population: Safety population
Measure: Number; unit: Treatment related AEs
Arm/Group | Azzalure Alone as Initial Treatment | Filler Alone as Initial Treatment
Number analyzed (Participants) | 29 | 31
Treatment related AEs | 36 | 26

ADVERSE EVENTS:
Groups:
- Group A (Azzalure): After Single Treatment: Group A received Azzalure alone as initial single treatment, and thereafter two combined treatments. Events reported in this section occurred after the single treatment was given but before the 1st combined treatment was given.
- Group B (Filler): After Single Treatment: Group B received filler alone as initial single treatment, and thereafter two combined treatments. Events reported in this section occurred after the single treatment was given but before the 1st combined treatment was given.
- Group A: After 1st Combined Treatment: Group A received Azzalure alone as initial single treatment, and thereafter two combined treatments. Events reported in this section occurred after the 1st combined treatment was given.
- Group B: After 1st Combined Treatment: Group B received filler alone as initial single treatment, and thereafter two combined treatments. Events reported in this section occurred after the 1st combined treatment was given.
- Group A: After 2nd Combined Treatment: Group A received Azzalure alone as initial single treatment, and thereafter two combined treatments. Events reported in this section occurred after the 2nd combined treatment was given.
- Group B: After 2nd Combined Treatment: Group B received filler alone as initial single treatment, and thereafter two combined treatments.Events reported in this section occurred after the 2nd combined treatment was given.
Arm/Group | Group A (Azzalure): After Single Treatment | Group B (Filler): After Single Treatment | Group A: After 1st Combined Treatment | Group B: After 1st Combined Treatment | Group A: After 2nd Combined Treatment | Group B: After 2nd Combined Treatment
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/31 | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/29 | 4/31 | 15/28 | 13/28 | 9/28 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Azzalure): After Single Treatment (N=29) | Group B (Filler): After Single Treatment (N=31) | Group A: After 1st Combined Treatment (N=28) | Group B: After 1st Combined Treatment (N=28) | Group A: After 2nd Combined Treatment (N=28) | Group B: After 2nd Combined Treatment (N=28)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Azzalure): After Single Treatment (N=29) | Group B (Filler): After Single Treatment (N=31) | Group A: After 1st Combined Treatment (N=28) | Group B: After 1st Combined Treatment (N=28) | Group A: After 2nd Combined Treatment (N=28) | Group B: After 2nd Combined Treatment (N=28)
Implant site bruising (General disorders) | 0 (0) | 0 (0) | 7 (14) | 4 (8) | 5 (8) | 4 (6)
Implant site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
VII nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haematoma (General disorders) | 0 (0) | 1 (2) | 3 (5) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Inflammatory reaction (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Lump (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephritic colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Redness
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes